CLINICAL TRIAL: NCT03604497
Title: Using Bluetooth Beacon Technology to Reduce Distracted Pedestrian Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, David Schwebel, Primary Investigator, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: R21HD095270 (NIH); R21HD095270 (NIH)
Record Dates: First submitted 2018-07-11; First posted 2018-07-27 (Actual); Results first posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- beacon alerts (Experimental): active intervention - participants are receiving alerts to warn them about distracted pedestrian behavior near intersections
  Interventions: Behavioral: beacon alerts
- no alerts baseline (No Intervention): baseline - participants do not receive any alerts on their mobile smartphone when near intersections
- no alerts retention (Other): retention phase - alerts have stopped after active intervention and behavior is monitored to test retention of learned behavior
  Interventions: Behavioral: no alerts retention

INTERVENTIONS:
Behavioral: beacon alerts — alerts via unidirectional communication from beacons to smartphones when smartphones are approaching pedestrian crossing at activated intersection
  Arms: beacon alerts
Behavioral: no alerts retention — no alerts will appear, but we will measure retention of behavior learned during the active intervention stage
  Arms: no alerts retention

SUMMARY:
Over 4,800 American pedestrians die annually, a figure that is current increasing. One hypothesized reason for the increasing trend in pedestrian injuries and deaths is the role of mobile technology in distracting both pedestrians and drivers. The investigators propose to develop and then evaluate Bluetooth beacon technology as a means to alert and warn pedestrians when they are approaching dangerous intersections, reminding them to attend to the traffic environment and cross the street safely rather than engaging with mobile technology. One aspect of the research will involve a crossover research trial to evaluate efficacy of the program.

Bluetooth beacons are very small (about the size of a dime) and inexpensive (~$20 range) devices that broadcast information unidirectionally (beacon to smartphone) within a closed proximal network. The investigators propose placing beacons at intersection corners (e.g., on signposts) frequently trafficked by urban college students. The beacons will transmit to an app installed on users' smartphones, signaling users to attend to their environment and cross the street safely. The app will be developed to be flexible based on user preferences; for research purposes, the app also will download data concerning the users' behavior while crossing the street. The crossover trial will evaluate the app with a sample of about 411 young adults whose behavior is monitored for: (a) 3 weeks without the app being activated, (b) 3 weeks with the app activated, and then (c) 6 weeks without the app activated to assess retention of behavior. Throughout the 12 week period, the investigators will monitor user behavior at multiple intersections around campus, along with gathering self-report questionnaire perceptions and behavior at baseline and 12-week post-intervention assessments.

ELIGIBILITY:
Inclusion Criteria:

* individuals who cross streets on the UAB campus at least twice daily
* ownership of an Android phone
* willingness to install the app on phone
* ability to communicate in English

Exclusion Criteria:

* none

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 437 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2019-12-21 (Actual); Study Completion 2019-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C Schwebel, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Youth Safety Lab, University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Will communicate with qualified investigators to share anonymous data if research goals are justified
Supporting Information: Study Protocol, ICF
Time Frame: after publication of final results and for 3 years
Access Criteria: contact study PI

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 437 individuals enrolled and 385 crossed the street at least once during the protocol, suggesting they participated. The numbers do not add up since it is a crossover trial.
Groups:
- All Study Participants: baseline - participants do not receive any alerts on their mobile smartphone when near intersections
  active intervention phase - participants are receiving alerts to warn them about distracted pedestrian behavior near intersections (beacon alerts: alerts via unidirectional communication from beacons to smartphones when smartphones are approaching pedestrian crossing at activated intersection)
  retention phase - alerts have stopped after active intervention and behavior is monitored to test retention of learned behavior (no alerts retention: no alerts will appear, but we will measure retention of behavior learned during the active intervention stage)
  All participants engaged in all three phrases in the same order
Period: Overall Study
Arm/Group | All Study Participants
Started | 437
Completed | 385
Not Completed | 52
Not completed — Protocol Violation | 52

BASELINE CHARACTERISTICS:
Population: Analysis population is same as assignment in participant flow.
Groups:
- All Study Participants: baseline - participants do not receive any alerts on their mobile smartphone when near intersections
  active intervention - participants are receiving alerts to warn them about distracted pedestrian behavior near intersections (beacon alerts: alerts via unidirectional communication from beacons to smartphones when smartphones are approaching pedestrian crossing at activated intersection)
  retention phase - alerts have stopped after active intervention and behavior is monitored to test retention of learned behavior (no alerts retention: no alerts will appear, but we will measure retention of behavior learned during the active intervention stage)
Arm/Group | All Study Participants
Number analyzed (Participants) | 437
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.2 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: A handful of participants declined to provide gender or indicated non-binary gender. Those cells are left as missing.
  Participants
    number analyzed (Participants) | 431
    Female | 287
    Male | 144
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/Black | 117
  Asian/Pacific Islander | 88
  Hispanic | 25
  Native American/American Indian/Alaskan Native | 4
  White | 178
  Other/Biracial/Biethnic/Prefer not to respond | 25
Region of Enrollment [Number; unit: participants]
  United States | 437

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Street Crossings Distracted
Description: percentage of street-crossings participants is distracted while crossing streets in intersections involved in the study, as measured electronically by smartphone behavior near those intersections. Electronic measurement was based on x-y-z coordinates of the smartphone during the crossing, as assessed and stored in the participants' phone storage.
Time Frame: 12 weeks
Population: Participants who crossed the street at least once during study protocol; crossover trial and all participants completed phases in the same order with no alerts baseline first, beacon alerts second, and no alerts retention third
Measure: Number; unit: per cent of crossings distracted
Arm/Group | Beacon Alerts | no Alerts Baseline | no Alerts Retention
Number analyzed (Participants) | 385 | 385 | 385
per cent of crossings distracted | 75 | 74 | 74

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Beacon Alerts | no Alerts Baseline | no Alerts Retention
All-Cause Mortality (participants affected / at risk) | 0/385 | 0/385 | 0/385
Serious Adverse Events (participants affected / at risk) | 0/385 | 0/385 | 0/385
Other Adverse Events (participants affected / at risk) | 0/385 | 0/385 | 0/385

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-08-16): https://cdn.clinicaltrials.gov/large-docs/97/NCT03604497/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-09): https://cdn.clinicaltrials.gov/large-docs/97/NCT03604497/SAP_001.pdf